CLINICAL TRIAL: NCT04731064
Title: Recurrence Rate of Hemorrhoidal Disease at 10 Years and More After Hemorrhoidal Artery Ligation (HAL)
Brief Title: Recurrence Rate of Hemorrhoidal Disease at 10 Years and More After HAL Doppler or HAL-RAR Intervention
Acronym: HALTY
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.283
Record Dates: First submitted 2021-01-28; First posted 2021-01-29 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Hemorrhoidal Disease
MeSH Terms: interventions — Retinoic Acid Receptor alpha

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: HAL (Hemorrhoidal Artery Ligation) - RAR (Recto-Anal Repair) — The patient is operated on in the first perineal position, under general anesthesia or under locoregional or even local anesthesia, after rectal preparation by simple enema. The HAL equipment included a disposable transparent rectoscope fitted near its end with a centimeter window through which wire stitch ligatures will be made. A light source facilitating the exposure of the internal face of the rectum and a Doppler transducer secured to the base of the rectoscope containing the Doppler system. Everything is connected to a generator which transmits Doppler noises to the surgeon. A printer on the generator makes it possible to map ligatures and note the depth of linked arteries. Equipment includes needle holder, knot pusher, scissors and dissecting forceps. The material for HAL is identical, except for the disposable rectoscope which is more indented at its end and on one side.

SUMMARY:
The treatment of hemorrhoidal disease involves both instrumental and surgical techniques (hemorrhoidectomy and hemorrhoidopexy). In 1995, a Japanese author proposed a new treatment technique for stage II (spontaneous reintegration prolapse) or III (digital reintegration prolapse) disease, based on Doppler identification of low perirectal arteries followed by their ligation, via a specific windowed rectoscope. Later, a further modification appeared, allowing patients to be treated at more advanced stages, adding vertical mucopexy to the ligatures along the main bundles.

The pathophysiology of hemorrhoidal disease is based on a vascular theory (opening of arteriovenous shunts) and on a mechanical theory (distension of the supporting tissue). Hemorrhoidectomy responds to the first, hemorrhoidopexy to the second. The HAL (Hemorrhoidal Artery Ligation) - RAR (Recto-Anal Repair) technique seeks to treat both vascular (by ligation of the nourishing arteries) and mechanical (by mucopexy of prolapsed bundles) components. The technique first spread to Germany, Russia, Italy, Spain, Australia and England. It has been popularized in France by some authors.

DETAILED DESCRIPTION:
The treatment of hemorrhoidal disease involves both instrumental and surgical techniques (hemorrhoidectomy and hemorrhoidopexy). In 1995, a Japanese author proposed a new treatment technique for stage II (spontaneous reintegration prolapse) or III (digital reintegration prolapse) disease, based on Doppler identification of low perirectal arteries followed by their ligation, by a specific windowed rectoscope. Later, a further modification appeared, allowing patients to be treated at more advanced stages, adding vertical mucopexy to the ligatures along the main bundles.

Physiopathological basis of HAL Doppler The pathophysiology of hemorrhoidal disease is based on a vascular theory (opening of arteriovenous shunts) and on a mechanical theory (distension of the supporting tissue). Hemorrhoidectomy responds to the first, hemorrhoidopexy to the second. The HAL (Hemorrhoidal Arttery Ligation) - RAR (Recto-Anal Repair) technique seeks to treat both vascular components (by ligation of the nourishing arteries) and mechanical (by mucopexy of prolapsed bundles). The technique first spread to Germany, Russia, Italy, Spain, Australia and England. It was popularized in France by some authors.

Description of the operation The patient is operated on in the perineal first position, under general anesthesia or under locoregional or even local anesthesia. Most of the time, the procedure is performed on an outpatient basis, after rectal preparation with a simple enema.4,5 The equipment (there are several types) for HAL comprises a transparent disposable rectoscope provided near its end with a centimeter window through which the x-point ligatures of slowly absorbable 2/0 thread will be made. It contains a light source facilitating the exposure of the internal surface of the rectum and a Doppler transducer secured to the base of the rectoscope containing the Doppler system itself. The assembly is connected to a generator which will transmit the Doppler noises to the surgeon. A printer on the generator allows ligatures to be mapped and the depth of linked arteries to be noted.6 The rest of the equipment includes a needle holder, knot pusher, scissors and dissecting forceps to dab the surgical site if necessary.2 The material for HAL with mucopexy is identical, except for the disposable rectoscope which is much more indented at its end and on one side (and at the time of arterial ligation, covered by a metal or opalescent jacket leaving a window), so as to be able to carry out a vertical overlock in the lower rectum, above the package that the operator intends to treat. It is thus possible to make one or more mucopexies depending on the operative findings.

The procedure takes about 20 to 30 minutes. Two circumferential explorations are performed at the level of the lower rectum, approximately 25 and 40 mm above the pectinate line. Patients on anticoagulant or antiplatelet therapy can be operated using this technique, since there is no wound. The patient leaves the same day with paracetamol on demand, without special care at home.

ELIGIBILITY:
Inclusion Criteria:

* Patient operated for hemorrhoidal disease for 10 or more
* Age 18 and over
* Informed patients

Exclusion Criteria:

* Patient opposition
* Minor patient

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients operated for a disease in the digestive surgery and emergency departments will be included, provided they are not opposed.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The rate of recurrence leading to a re-intervention within 10 years of the intervention. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Giorgia Mastronicola, Principal Investigator — CHU Grenoble Alpes; Jean Luc FAUCHERON, MD-PhD, Study Director — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble-alpes, Grenoble, France